CLINICAL TRIAL: NCT01194895
Title: Impact of Intraoperative Protective One-lung Ventilation in Patients Undergoing Esophagectomy : a Prospective Randomized Controlled Trial
Brief Title: A Trial to Evaluate the Impact of Lung-protective Intervention in Patients Undergoing Esophageal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Ming Zhong, department of anesthesiology and surgical intensive care unit, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ESO-2010-LV; ESOPV (Other: SICU)
Record Dates: First submitted 2010-08-18; First posted 2010-09-03 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Acute Lung Injury
Keywords: esophagectomy; acute lung injury; protective ventilation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- protective ventilation (Experimental)
  Interventions: Other: protective ventilation
- conventional ventilation (Active Comparator)
  Interventions: Other: conventional ventilation

INTERVENTIONS:
Other: protective ventilation — set tidal volume of 5ml/kg during one-lung ventilation
  Other Names: low tidal volume ventilation
  Arms: protective ventilation
Other: conventional ventilation — keep tidal volume at 8ml/kg during one-lung ventilation
  Other Names: normal tidal volume ventilation
  Arms: conventional ventilation

SUMMARY:
The purpose of this trial is to determine whether low tidal volume during intraoperative one-lung ventilation could decrease the incidence rate of postoperative acute lung injury compared to "normal" tidal volume.

DETAILED DESCRIPTION:
Large tidal volume are known risk factor of acute lung injury.Mechanical ventilation with low tidal volume has been shown to attenuate lung injuries in critically ill patients.Esophagectomy surgery need a relatively long time of one-lung ventilation. A normal tidal volume of two-lung ventilation should be a large one when exerted to one lung. We hypothesized that low tidal volume ventilation during one-lung ventilation could decrease incidence rate of postoperative acute lung injury and mortality.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of esophageal carcinoma and planned for esophagectomy
* indication for one-lung ventilation
* informed consent
* ASA I~II

Exclusion Criteria:

* NYHA III~IV
* severe COPD
* pulmonary fibrosis
* any new pulmonary infiltrate on chest radiograph
* preoperative acute infection suspected
* altered liver function( Child-Pugh class B or moe)
* acute or chronic renal failure
* preoperative corticosteroid treatment during month before inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
cytokines of bronchoalveolar lavage | 10 minutes before surgery ,at the end of surgery immediately
  TNF-a,IL-1b,IL-6,IL-8 of BAL will be measured with enzyme-linked immunoassay,all markers will be reported with a unit of pg/ml

SECONDARY OUTCOMES:
postoperative hospital days | after surgery up to the time when patient is discharged or dead，it is an average
  duration of hospital stay after surgery
incidence rate of acute lung injury | after surgery up to 28 days
  Diagnosis of acute lung injury is followed the consensus criteria for ALI/ARDS published in "Am J Respir Crit Care Med 1994, 149:818-824".
incidence rate of surgical complications | after surgery up to 28 days
  surgical complications include anastomotic fistula, postoperative infection and the patients will be followed until death or discharged
inhospital mortality | after surgery up to 28 days
  the number of death in the period of hospital stay
Oxygenation Index | 10 minutes before surgery,at the end of surgery immediately,12h after surgery
  Oxygenation Index=PaO2/FiO2
CT scan of chest | 12 hours after the surgery
  Severity of pulmonary edema will be evaluated by CT scan of chest

CONTACTS AND LOCATIONS:
Overall Officials: Zhanggang Xue, professor, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, China

REFERENCES:
- [Derived] Shen Y, Zhong M, Wu W, Wang H, Feng M, Tan L, Wang Q. The impact of tidal volume on pulmonary complications following minimally invasive esophagectomy: a randomized and controlled study. J Thorac Cardiovasc Surg. 2013 Nov;146(5):1267-73; discussion 1273-4. doi: 10.1016/j.jtcvs.2013.06.043. Epub 2013 Aug 28. PMID 23993028